CLINICAL TRIAL: NCT06897605
Title: Clinical Study Evaluating the Impact of Dapagliflozin on Erythropoiesis-Stimulating Agent Responsiveness in Anemic Patients With Chronic Kidney Disease
Brief Title: Impact of Dapagliflozin in Anemic Chronic Kidney Disease Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Principal investigator-Associate Professor of Clinical Pharmacy-Clinical Pharmacy and Pharmacy Practice Department, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-117'1
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease(CKD); Anemia, Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia; Kidney Diseases; Bronchiolitis Obliterans Syndrome | interventions — dapagliflozin; Hematinics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin + ESA group (Experimental): patients will receive dapagliflozin 10 mg tablet once daily in addition to standard care therapy of erythropoiesis-stimulating agents (ESA)
  Interventions: Drug: Dapagliflozin (DAPA); Drug: Erythropoiesis Stimulating Agent
- Control group (Other): patients will receive standard care therapy of erythropoiesis-stimulating agents (ESA)
  Interventions: Drug: Erythropoiesis Stimulating Agent

INTERVENTIONS:
Drug: Dapagliflozin (DAPA) — Dapagliflizin 10 mg tablets once daily for 12 weeks
  Arms: Dapagliflozin + ESA group
Drug: Erythropoiesis Stimulating Agent — Erythropoiesis stimulating agent (ESA) therapy

SUMMARY:
Dapagliflozin is a sodium-glucose co-transporter 2 (SGLT2) inhibitor, primarily used in the management of type 2 diabetes mellitus. Emerging research suggests that SGLT2 inhibitors may offer additional benefits, including reducing the risk of cardiovascular events and renal complications. Post hoc analyses of previous clinical trials have shown that patients treated with SGLT2 inhibitors exhibited higher levels of hemoglobin and hematocrit compared to those in the control group. These findings suggest that dapagliflozin's ability to elevate hemoglobin levels could potentially be utilized for the treatment of anemia in patients with chronic kidney disease.

ELIGIBILITY:
Inclusion criteria

1. Adults aged ≥ 18 years with CKD stage III or IV.
2. Patients with anemia of CKD and a hemoglobin level < 11.5 g/dL
3. Patients are receiving erythropoiesis-stimulating agent therapy.

Exclusion criteria

1. Anemia due to causes other than chronic kidney disease, such as pernicious anemia, thalassemia, sickle cell anemia, or myelodysplastic syndromes.
2. Patients with severe ketosis, diabetic coma, severe infection, perioperative complications, or severe trauma.
3. Patients with acute heart failure, acute myocardial infarction, or stroke occurring within 6 months before enrollment in the trial.
4. Patients with current malignancies or a history of malignancy within the past 2 years.
5. Diagnosed with pure red cell aplasia.
6. Patients with severe gastrointestinal bleeding.
7. Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in Erythropoiesis stimulating agent therapy dose | 12 weeks
  Difference between two groups in comulative dose of erythropoiesis stimulating agent therapy (E.S.A) in international unit (I.U) at the end of the study.

SECONDARY OUTCOMES:
Changes in hemoglobin level | 12 weeks
  Difference between two groups in hemoglobin level in g/dL at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Noha O. Mansour, Ph.D., Principal Investigator — Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Egypt